CLINICAL TRIAL: NCT00002254
Title: A Multi-Center, Open-Label, Ascending, Multiple Oral Dose, Safety, Tolerance and Pharmacokinetic Study of 3'-Deoxy-3'-Fluorothymidine (FLT) in Patients With Acquired Immune Deficiency Syndrome (AIDS) or AIDS-Related Complex (ARC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lederle Laboratories (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 054B; 81-2
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-05

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — alovudine

INTERVENTIONS:
Drug: Alovudine

SUMMARY:
To assess the tolerance and toxicity profile of deoxy-3'-fluorothymidine (FLT) after multiple oral dosing for 16 weeks. To characterize the steady-state pharmacokinetics of FLT after multiple oral doses. To assess the effect of FLT on immunologic and virologic markers of HIV infection (CD4+ lymphocyte count, p24 antigen, viremia) in patients with AIDS or AIDS related complex (ARC) after multiple oral dosing for 16 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aerosolized pentamidine for Pneumocystis carinii pneumonia (PCP) prophylaxis.
* Up to 14 days of systemic therapy for minor opportunistic infections such as candidiasis, mucocutaneous Herpes simplex or cutaneous Herpes zoster infections.

Patients must have the following:

* AIDS or AIDS related complex (ARC) as defined by the CDC.
* Positive antibody to HIV as determined by a commercially licensed ELISA test kit, confirmed by Western blot analysis.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Symptomatic visceral Kaposi's sarcoma or progression of Kaposi's sarcoma within the month prior to study entry (progression is defined as more than a 25 percent increase in the product of bidirectional measurement of indicator lesions and/or more than a 25 percent increase in the number of new lesions).
* Concurrent neoplasms other than Kaposi's sarcoma or basal cell carcinoma of the skin. Patients who have had a malignancy in the past that has been in complete remission for 1 year without therapy may be enrolled.
* Signs or symptoms of neuropathy and a Vibratron 2 score = or > 4 for either great toe.

Concurrent Medication:

Excluded:

* Acute therapy for AIDS-related infection.
* Systemic maintenance therapy for AIDS-defining opportunistic infection.
* Recombinant erythropoietin.
* Long term therapy with either aspirin or probenecid.

Concurrent Treatment:

Excluded:

* Blood transfusion more than once per month.

Patients with the following are excluded:

* Symptomatic visceral Kaposi's sarcoma or progression of Kaposi's sarcoma within the month prior to study entry.
* Unwilling to sign an informed consent or patients unwilling to be followed at the medical center where they were enrolled for the duration of the study and follow-up as required.
* History of intolerance to zidovudine (AZT) at any dose as demonstrated by an AZT related decrease in hemoglobin levels of at least 2 g/dl or AZT related depression of neutrophils of at least 200 cells/mm3 to < 750 cells/mm3 which required discontinuation of AZT therapy.
* Diseases or conditions listed in Exclusion Co-Existing Conditions.

Prior Medication:

Excluded:

* Antiretroviral agents within 14 days of study entry.
* Immunomodulating agents or corticosteroids within 30 days prior to study entry.
* Treatment for acute Pneumocystis carinii pneumonia within 2 weeks prior to study entry.

Prior Treatment:

Excluded:

* Blood transfusions within 7 days prior to study entry.
* Radiation therapy for Kaposi's sarcoma within 30 days prior to study entry.

Active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Univ of North Carolina School of Medicine, Chapel Hill, North Carolina

REFERENCES:
- [Background] Barditch-Crovo PA, Kornhauser DM, Petty BG, Nerhood LJ, Lietman PS, Faulkner R, Ganes D, Kuye O, Flexner C. Phase I pharmacokinetic evaluation of 3'deoxy-3'-fluorothymidine (FLT), a new potent anti-HIV nucleoside. Int Conf AIDS. 1991 Jun 16-21;7(2):210 (abstract no WB2114)